CLINICAL TRIAL: NCT01343147
Title: Deep Versus Superficial Heating in Patients With Knee Osteoarthritis: a Double-blind Randomized Clinical Trial
Brief Title: Deep Versus Superficial Heating in Patients With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Carlo Bertolini, Principal Investigator, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 533/10
Record Dates: First submitted 2011-04-26; First posted 2011-04-27 (Estimated); Last update posted 2014-03-05 (Estimated); Status verified 2014-03

CONDITIONS: Knee Osteoarthritis
Keywords: Hyperthermia; Microwave diathermy; Hot packs; Pain; Physical function
MeSH Terms: conditions — Osteoarthritis, Knee; Hyperthermia; Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Deep hyperthermia (Other): Microwave diathermy
  Interventions: Other: Microwave diathermy
- Superficial hyperthermia (Other): Hot packs
  Interventions: Other: Superficial hyperthermia

INTERVENTIONS:
Other: Microwave diathermy — Deep tissue heating via microwave diathermy
  Arms: Deep hyperthermia
Other: Superficial hyperthermia — Superficial heating via hot pack application
  Arms: Superficial hyperthermia

SUMMARY:
Heat therapy is frequently prescribed to patients with symptomatic knee osteoarthritis (OA). Deep hyperthermia via localized microwave diathermy is effective in several musculoskeletal painful conditions. However, the efficacy of superficial heating is controversial. Furthermore, no clinical trials have yet directly compared the effects of these treatment modalities in knee OA. Hence, the purpose of the present study is to compare the effects of deep and superficial hyperthermia, induced via microwave diathermy and hot packs, respectively, on pain and function in patients with symptomatic knee OA.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 years or older
* Moderate, mono or bilateral knee osteoarthritis
* Pain lasting for at least three weeks

Exclusion Criteria:

* Inability or unwillingness to sign informed consent
* Previous surgery on the affected knee
* Intra-articular injections with steroids or hyaluronic acid in prior 6 months
* Physical therapy for knee problems in prior 6 months
* Congenital or acquired inflammatory or neurological (systemic or local) diseases involving the knee
* Chronic NSAID or steroid treatment
* Cognitive or psychiatric disorders
* Pregnancy or breastfeeding
* Contraindications to hyperthermia (cancer in prior 2 years or active cancer treatment, local thrombosis, impaired arterial circulation, altered cutaneous thermal sensitivity, local infections or systemic acute infections, metal implants or prosthesis, severe osteoporosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2010-05; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC scale) | 12 months

SECONDARY OUTCOMES:
British Medical Research Council (BMRC) rating scale | 6 months
Pain visual analogue scale (VAS) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Bertolini, M.D., Principal Investigator — Catholic University of the Sacred Heart
Locations (1):
- Outpatient clinic of the Dept. Of Gerontology, Geriatrics and Physiatrics, Rome, Italy

REFERENCES:
- [Background] Giombini A, Giovannini V, Di Cesare A, Pacetti P, Ichinoseki-Sekine N, Shiraishi M, Naito H, Maffulli N. Hyperthermia induced by microwave diathermy in the management of muscle and tendon injuries. Br Med Bull. 2007;83:379-96. doi: 10.1093/bmb/ldm020. PMID 17942453
- [Background] Di Cesare A, Giombini A, Dragoni S, Agnello L, Ripani M, Saraceni VM, Maffulli N. Calcific tendinopathy of the rotator cuff. Conservative management with 434 Mhz local microwave diathermy (hyperthermia): a case study. Disabil Rehabil. 2008;30(20-22):1578-83. doi: 10.1080/09638280701786351. PMID 18608369
- [Background] Giombini A, Di Cesare A, Safran MR, Ciatti R, Maffulli N. Short-term effectiveness of hyperthermia for supraspinatus tendinopathy in athletes: a short-term randomized controlled study. Am J Sports Med. 2006 Aug;34(8):1247-53. doi: 10.1177/0363546506287827. Epub 2006 Apr 24. PMID 16636345
- [Background] Kaplan LD, Chu CR, Bradley JP, Fu FH, Studer RK. Recovery of chondrocyte metabolic activity after thermal exposure. Am J Sports Med. 2003 May-Jun;31(3):392-8. doi: 10.1177/03635465030310031101. PMID 12750132
- [Background] Weinberger A, Fadilah R, Lev A, Levi A, Pinkhas J. Deep heat in the treatment of inflammatory joint disease. Med Hypotheses. 1988 Apr;25(4):231-3. doi: 10.1016/0306-9877(88)90036-9. PMID 3367814
- [Background] Cetin N, Aytar A, Atalay A, Akman MN. Comparing hot pack, short-wave diathermy, ultrasound, and TENS on isokinetic strength, pain, and functional status of women with osteoarthritic knees: a single-blind, randomized, controlled trial. Am J Phys Med Rehabil. 2008 Jun;87(6):443-51. doi: 10.1097/PHM.0b013e318174e467. PMID 18496246
- [Background] Robertson VJ, Ward AR, Jung P. The effect of heat on tissue extensibility: a comparison of deep and superficial heating. Arch Phys Med Rehabil. 2005 Apr;86(4):819-25. doi: 10.1016/j.apmr.2004.07.353. PMID 15827938